CLINICAL TRIAL: NCT00693680
Title: The Role of Zinc in Therapy of Unipolar Depression
Brief Title: Zinc Supplementation of Imipramine Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Polish Academy of Sciences (Other)
Collaborators: Jagiellonian University (Other)
Responsible Party: prof. Gabriel Nowak, Institute of Pharmacology, Polish Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZnIMI/2004
Record Dates: First submitted 2008-06-05; First posted 2008-06-09 (Estimated); Last update posted 2008-06-13 (Estimated); Status verified 2008-06

CONDITIONS: Major Depression
Keywords: depression; antidepressant treatment; zinc; placebo
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Imipramine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): zinc + imipramine
  Interventions: Dietary Supplement: Zincas Forte
- 2 (Placebo Comparator): placebo + imipramine
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Zincas Forte — 25 mgZn/day + imipramine (100-200mg/day)
  Other Names: Zincas Forte (Farmapol, Poland); Imipramin (Polfarma, Poland)
  Arms: 1
Dietary Supplement: Placebo — placebo + imipramine (100-200mg/day)
  Other Names: Imipramin (Polfarma, Poland)
  Arms: 2

SUMMARY:
Examination of the effect of zinc supplementation on imipramine therapy in major depression.

DETAILED DESCRIPTION:
A placebo-controlled, double blind study of zinc supplementation in imipramine therapy was conducted in sixty, depressed patients fulfilling the DSM-IV criteria for major depression without psychotic symptoms. After a one week washout period, patients were randomized into two groups treated with imipramine and receiving once daily either placebo (n=30) or zinc supplementation (n=30) for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* patients with fulfilled DSM-IV criteria for moderate or severe depressive episode
* one week washout period without any pharmacotherapy

Exclusion Criteria:

* psychotic symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-01; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
To compare the effect of zinc vs placebo in imipramine treated depressed patients (CGI, BDI, HADRS, MADRS) | 12 weeks

SECONDARY OUTCOMES:
To assess unwanted side effects in both groups | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Zieba, Prof., Principal Investigator — Department of Psychiatry, Collegium Medicum
Locations (1):
- Department of Psychiatry, Collegium Medicum, Jagiellonian University, Krakow, Poland

REFERENCES:
- [Background] Nowak G, Siwek M, Dudek D, Zieba A, Pilc A. Effect of zinc supplementation on antidepressant therapy in unipolar depression: a preliminary placebo-controlled study. Pol J Pharmacol. 2003 Nov-Dec;55(6):1143-7. PMID 14730113